CLINICAL TRIAL: NCT06661226
Title: Comparative Effects of Acceleration Drills and Change in Direction Drills on Agility, Speed and Performance in Squash Players
Brief Title: Acceleration Drills and Change in Direction Drills on Agility, Speed and Performance in Squash Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0408
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Sports Physical Therapy
Keywords: Acceleration Drills; Agility Training; Change in Direction Drills; Squash

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceleration Drills (Experimental): 14 participants will be in experimental group A, giving them acceleration drill protocol for six weeks. Measure all values before giving them protocol and after protocol.
  Interventions: Other: Accleration drills
- Change in Direction Drills (Experimental): 14 participants will be in experimental group B, giving them Change in direction drill protocol for six weeks. Measure all values before giving them protocol and after protocol.
  Interventions: Other: Change in Direction Drills

INTERVENTIONS:
Other: Accleration drills — 14 participants will be in experimental group A, giving them acceleration drill protocol for six weeks. Measure all values before giving them protocol and after protocol.
  Arms: Acceleration Drills
Other: Change in Direction Drills — 14 participants will be in experimental group B, giving them Change in direction drill protocol for six weeks. Measure all values before giving them protocol and after protocol.
  Arms: Change in Direction Drills

SUMMARY:
Squash match play is characterized by fast and frenetic movements, making the development of agility and speed crucial for players. The majority of movements in squash involve only 2 or 3 steps, emphasizing the need for quick and explosive movement execution.

It is a randomized clinical trial with non-probability convenience sampling technique. The sample size of the study is 28. It will be conducted in Punjab Squash Association in Lahore within 6 months after approval of synopsis. Group A will receive acceleration drills in 15-minute sessions for 6 weeks. 3-5 days per week with moderate to high intensity. Group B will receive change in direction drills (15-minute sessions) for 6 weeks, 3-5 times a week, with moderate to high intensity. The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 25.0. If data will be normally distributed, then parametric; if not normally distributed, then non-parametric.

The aim of the study is to compare the effects of acceleration drills versus change in direction drills on agility, speed, and performance in squash players.

DETAILED DESCRIPTION:
The objective of my study is to determine comparative effects of acceleration drills and change in direction drills on agility, speed, and performance in squash players.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 30.
* Only male players will be included.
* Players actively playing from last one year.
* Consistent play at a B/C or higher league level (adjust based on local/national ranking system)

Exclusion Criteria:

* Non-athletic population.
* History of recent injuries or medical conditions that would contra-indicate training.
* Players with any musculoskeletal injury.
* Players with any spine related issues.
* Players with shoulder pathology.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Illinois agility test | Time Frame 6 weeks
  Illinois agility test is used to test running agility using various turns and movements Participants should lie on their front and hands by their shoulders. On the 'Go' command, the stopwatch is started, and the athlete gets up as quickly as possible and runs forwards ten meters to run around a cone, then back ten meters, then runs up and back through a slalom course of four cones. Finally, the athlete runs another ten meters up and back past the finishing cone, at which the timing is stopped.
Sprint for speed | Time Frame 6 weeks
  The twenty meter sprint test used to evaluate the sprints. This test starts from the starting line with a standing position. Participants ran twenty meters as fast as possible. Time is evaluated for five, ten, fifteen and twenty meters. Record time in seconds. The faster the time, the better the speed.
Vertical jump test | Time Frame 6 weeks
  It is a standard test for measuring athletic performance. The athlete stands side on to a wall and reaches up with the hand closest to the wall. Keeping the feet flat on the ground, the point of the fingertips is marked or recorded. This is called the standing reach height. The athlete then stands away from the wall, and leaps vertically as high as possible using both arms and legs to assist in projecting the body upwards. Attempt to touch the wall at the highest point of the jump. The difference in distance between the standing reach height and the jump height is the score. The best of three attempts is recorded.
Squat One-repetition maximum (1RM) Test | Time Frame 6 weeks
  The One-repetition maximum test is considered as the 'gold standard' for assessing the strength capacity of individuals in non-laboratory environments. One-repetition maximum is a measure of the maximal weight a subject can lift with one repetition.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Punjab Squash Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loturco I, A Pereira L, T Freitas T, E Alcaraz P, Zanetti V, Bishop C, Jeffreys I. Maximum acceleration performance of professional soccer players in linear sprints: Is there a direct connection with change-of-direction ability? PLoS One. 2019 May 14;14(5):e0216806. doi: 10.1371/journal.pone.0216806. eCollection 2019. PMID 31086386
- [Background] McBride JM, Blow D, Kirby TJ, Haines TL, Dayne AM, Triplett NT. Relationship between maximal squat strength and five, ten, and forty yard sprint times. J Strength Cond Res. 2009 Sep;23(6):1633-6. doi: 10.1519/JSC.0b013e3181b2b8aa. PMID 19675504
- [Background] Ziv G, Lidor R. Vertical jump in female and male basketball players--a review of observational and experimental studies. J Sci Med Sport. 2010 May;13(3):332-9. doi: 10.1016/j.jsams.2009.02.009. Epub 2009 May 13. PMID 19443269
- [Background] Williams BK, Sanders RH, Ryu JH, Graham-Smith P, Sinclair PJ. The kinematic differences between accurate and inaccurate squash forehand drives for athletes of different skill levels. J Sports Sci. 2020 May;38(10):1115-1123. doi: 10.1080/02640414.2020.1742971. Epub 2020 Mar 29. PMID 32223529
- [Background] Chandra S, Sharma A, Malhotra N, Rizvi MR, Kumari S. Effects of Plyometric Training on the Agility, Speed, and Explosive Power of Male Collegiate Badminton Players. J Lifestyle Med. 2023 Feb 28;13(1):52-58. doi: 10.15280/jlm.2023.13.1.52. PMID 37250280
- [Background] Gabbett TJ, Sheppard JM, Pritchard-Peschek KR, Leveritt MD, Aldred MJ. Influence of closed skill and open skill warm-ups on the performance of speed, change of direction speed, vertical jump, and reactive agility in team sport athletes. J Strength Cond Res. 2008 Sep;22(5):1413-5. doi: 10.1519/JSC.0b013e3181739ecd. PMID 18714250
- [Background] Paul DJ, Gabbett TJ, Nassis GP. Agility in Team Sports: Testing, Training and Factors Affecting Performance. Sports Med. 2016 Mar;46(3):421-42. doi: 10.1007/s40279-015-0428-2. PMID 26670456
- [Background] Lockie RG, Post BK, Dawes JJ. Physical Qualities Pertaining to Shorter and Longer Change-of-Direction Speed Test Performance in Men and Women. Sports (Basel). 2019 Feb 16;7(2):45. doi: 10.3390/sports7020045. PMID 30781530
- [Background] Girard O, Micallef JP, Noual J, Millet GP. Alteration of neuromuscular function in squash. J Sci Med Sport. 2010 Jan;13(1):172-7. doi: 10.1016/j.jsams.2008.11.002. Epub 2009 Feb 23. PMID 19231287
- [Background] James C, Dhawan A, Jones T, Pok C, Yeo V, Girard O. Minimal Agreement between Internal and External Training Load Metrics across a 2-wk Training Microcycle in Elite Squash. J Sports Sci Med. 2021 Mar 1;20(1):101-109. doi: 10.52082/jssm.2021.101. eCollection 2021 Mar. PMID 33707993
- [Background] James C, Jones T, Farra S. Physiological and Performance Correlates of Squash Physical Performance. J Sports Sci Med. 2022 Feb 15;21(1):82-90. doi: 10.52082/jssm.2022.82. eCollection 2022 Mar. PMID 35250337
- [Background] McKay AKA, Stellingwerff T, Smith ES, Martin DT, Mujika I, Goosey-Tolfrey VL, Sheppard J, Burke LM. Defining Training and Performance Caliber: A Participant Classification Framework. Int J Sports Physiol Perform. 2022 Feb 1;17(2):317-331. doi: 10.1123/ijspp.2021-0451. Epub 2022 Dec 29. PMID 34965513
- [Background] James C, Dhawan A, Jones T, Girard O. Quantifying Training Demands of a 2-Week In-Season Squash Microcycle. Int J Sports Physiol Perform. 2021 Jun 1;16(6):779-786. doi: 10.1123/ijspp.2020-0306. Epub 2021 Feb 4. PMID 33547264
- [Background] Fernandez-Fernandez J, Garcia-Tormo V, Santos-Rosa FJ, Teixeira AS, Nakamura FY, Granacher U, Sanz-Rivas D. The Effect of a Neuromuscular vs. Dynamic Warm-up on Physical Performance in Young Tennis Players. J Strength Cond Res. 2020 Oct;34(10):2776-2784. doi: 10.1519/JSC.0000000000003703. PMID 32986392
- [Background] Ventura Comes A, Sanchez-Oliver AJ, Martinez-Sanz JM, Dominguez R. Analysis of Nutritional Supplements Consumption by Squash Players. Nutrients. 2018 Sep 20;10(10):1341. doi: 10.3390/nu10101341. PMID 30241327
- [Background] Turner O, Mitchell N, Ruddock A, Purvis A, Ranchordas M. Elite squash players nutrition knowledge and influencing factors. J Int Soc Sports Nutr. 2021 Jun 10;18(1):46. doi: 10.1186/s12970-021-00443-3. PMID 34112186
- [Background] Zubac D, Paravlic A, Koren K, Felicita U, Simunic B. Plyometric exercise improves jumping performance and skeletal muscle contractile properties in seniors. J Musculoskelet Neuronal Interact. 2019 Mar 1;19(1):38-49. PMID 30839302